CLINICAL TRIAL: NCT02299661
Title: An Open-Label, Randomised, Parallel Group Pilot Study to Assess the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Single Doses of DS-1093a in Patients With Chronic Kidney Disease
Brief Title: Pilot PK/PD Study of DS-1093a in Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DS1093-A-E103; 2014-002331-33 (EudraCT Number)
Record Dates: First submitted 2014-11-18; First posted 2014-11-24 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2015-06

CONDITIONS: Chronic Renal Disease; Renal Anemia
Keywords: Hypoxia inducible factor prolyl hydroxylase inhibitor.; Erythropoietin stimulating agent; Chronic renal disease; renal anemia
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 7.5mg DS-1093a (Experimental): DS-1093a, single oral dose of 7.5 mg
  Interventions: Drug: DS-1093a
- 25mg DS-1093a (Experimental): DS-1093a, single oral dose of 25 mg
  Interventions: Drug: DS-1093a
- 50mg DS-1093a (Experimental): DS-1093a, single oral dose of 50 mg
  Interventions: Drug: DS-1093a

INTERVENTIONS:
Drug: DS-1093a — DS-1093a, single oral doses up to 50 mg

SUMMARY:
DS-1093a is an inhibitor of hypoxia-inducible factor prolyl hydroxylases, and is expected to produce transient dose / exposure dependent increases in erythropoietin levels in subjects with chronic kidney disease (CKD). This study will be conducted in 2 parts. Part A will involve subjects with stage 3b or 4 CKD, and will be an open, non-controlled parallel group investigation of three single doses of DS-1093a (6 subjects/dose), in which allocation to dose will be randomised. On completion of this part of the study an optional fourth dose may be tested to gain a more complete understanding of the PK/PD behaviour of DS-1093a. Part B will be an open, non-controlled investigation of a single dose of DS-1093a in CKD subjects (n=6) receiving haemodialysis. The dose for Part B will be determined based on the data from Part A.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 - 70 years (inclusive).
* Female patients must be of non-childbearing potential (post-menopause or surgical sterilization). In women younger than 60 years a follicle-stimulating hormone (FSH) test will be conducted to confirm post-menopausal status (i.e., FSH ≥ 30 mU/mL).
* Part A: CKD stage 3b (eGFR: < 45 to ≥ 30 mL/min) or stage 4 (eGFR: < 30 to ≥ 15 mL/min). The CKD-EPI equation will be used for the eGFR estimation.
* Part B: Patients on chronic haemodialysis for at least 6 months and stable Hb levels (i.e., +/- 1 g/dL) for the last 6 months.
* Patient can be washed out from ESAs for at least 3 weeks (2 weeks prior to dosing and 1 week post-dose).
* Baseline Hb level ≥10 g/dL.
* Willingness to give written consent to participate after reading the ICF, and after having the opportunity to discuss the trial with the Investigator or his delegate.
* Male patients must be willing to use a reliable method of contraception during the trial, and for 4 months afterwards

Exclusion Criteria:

* Use of ESAs within 2 weeks prior to dosing.
* Uncontrolled hypertension despite optimal medical therapy, defined as > 160/100 mmHg after 10 minutes of rest at screening, and > 180/110 mmHg after 10 minutes of rest on Day -1 pre-dose.
* Known haemoglobinopathy.
* Acute renal failure (as judged by the Investigator).
* History of kidney transplant regardless of functionality.
* Start of any new medication or any changes to a current dosage within 7 days prior to study drug administration.
* Chronic liver disease.
* Positive hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody test.
* Positive test for human immunodeficiency virus (HIV)-1 or HIV-2.
* A history of gastrointestinal bleeding.
* History of a thrombotic event (e.g., myocardial infarction, stroke or transient ischemic attack, peripheral embolism, venous thromboembolism, etc.)
* Patients with poorly controlled diabetes despite optimal medical therapy.
* A history of cancer, except basal cell skin cancer, squamous cell skin cancer, or cervical cancer (if judged by the Investigator to be in full remission).
* Hypersensitivity to any components of the study drug.
* Requirement for any concomitant medication that cannot be withheld on Day 1 until 4 hours post-dose (insulin is allowed to cover the breakfast, if necessary).
* Clinically relevant abnormal medical history, physical findings, ECG, or laboratory values at the screening assessments that could interfere with the objectives of the trial or the safety of the patient.
* Participation in another investigational drug trial within 30 days prior to dosing (or 5 times the half-life of the drug, whichever is longer) or exposure to more than three new investigational agents within 12 months prior to enrolment.
* Abuse of drugs or alcohol during the 2 years before the first dose of trial medication.
* Ingestion of alcohol within 72 hours prior to dosing and during confinement. Outside the in-house period, regular alcohol consumption must not exceed 16 units for males and 7 units for females per week (1 unit equals 340 mL of beer, 115 mL of wine or 43 mL of spirits).
* Positive drug screen (if not due to concomitant medication) or alcohol breath test at screening and/or Day -1.
* Patients who smoke more than 10 cigarettes per day (or equivalent), and who would not be able to abstain from smoking during the in-house period.
* Concomitant use of medications known to affect the elimination of serum creatinine (e.g., trimethoprim or cimetidine) and competitors of renal tubular secretion (e.g., probenecid) within 30 days before dosing.
* Use of a strong inducer or inhibitor of CYP enzymes, during the 30 days before dosing.
* Use of any other prohibited medication.
* Loss of more than 400 mL blood, or donation of blood, plasma, platelets, or any other blood components, during the 3 months before the trial, or unwilling to abstain from donating during the study and for 3 months after receipt of the final dose of trial medication.
* Possibility that the patient will not cooperate with the requirements of the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of DS-1093a | 28 days
  Plasma concentrations of DS-1093a and derived PK parameters up to 28 days post-dose.
Change in serum erythropoietin concentrations | 6 days
  Change in serum erythropoietin concentrations compared to baseline, and derived EPO parameters, up to 6 days post-dose

SECONDARY OUTCOMES:
Change from baseline for composite haematology parameters | 28 days
  Change from baseline for haematology parameters (reticulocyte count, haemoglobin concentration, haematocrit, red blood cell count) up to 28 days post-dose.
Change from baseline for composite iron metabolism parameters | 7 days
  Change from baseline for iron metabolism parameters (serum concentrations of iron, transferrin, transferrin saturation, hepcidin-25) up to 7 days post-dose.
Change from baseline for serum concentrations of vascular endothelial growth factor | 7 days
  Change from baseline for serum concentrations of vascular endothelial growth factor up to 7 days post-dose
Number and severity of adverse events | 28 days
  Safety and tolerability up to 28 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Mendel Jansen, BSc, Study Director — Daiichi Sankyo Development
Locations (3):
- Czechia (2):
  - : Hemodialysis Center, Teaching Hospital Hradec Králove, Hradec Králové
  - PRA Clinical Pharmacology Unit, Prague
- PRA Clinical Pharmacology Unit, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/